CLINICAL TRIAL: NCT05074160
Title: OCS Liver Perfusion (OLP) Post-Approval Registry
Status: Active, not recruiting | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCSLIVER-01-PAS
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- OLP Registry primary analysis population: Adult primary liver transplant recipients who are transplanted with an OCS perfused DBD or DCD donor liver according to the approved indication and matching eligibility criteria
  Interventions: Device: OCS Liver

INTERVENTIONS:
Device: OCS Liver — Multi-center, observational post-approval registry of adult primary liver transplant recipients who are transplanted with an OCS Liver-perfused DBD or DCD donor liver according to the approved indication and that match the eligibility criteria below.

SUMMARY:
The objective of the OLP Registry is to collect more data on the post-transplant clinical outcomes of DBD and DCD donor livers preserved and assessed on OCS Liver System according to the approved indication and the OCS device performance in the real-world setting.

DETAILED DESCRIPTION:
OLP Registry is a multi-center, observational post-approval registry of adult primary liver transplant recipients who are transplanted with an OCS Liver-perfused DBD or DCD donor liver according to the approved indication and that match the eligibility criteria below.

ELIGIBILITY:
Inclusion Criteria:

* Adult primary liver transplant recipients of DBD or DCD donor Livers perfused on OCS Liver System

Donor Exclusion Criteria:

* Donor livers with accessory arterial blood supply requiring back table anastomosis, major traumatic injury, or hematoma; or
* Split donor liver; or
* DCD donor liver with >30 minutes of warm ischemic time (defined as from withdrawal of life support until donor liver cold flush); or
* DCD donors age >55 years; or
* DCD donor liver with macrosteatosis of >15%
* Living donors
* Donors with positive serology for HIV, Hep B and C
* Donors with macrosteatosis of ≥40%

Recipient Exclusion Criteria:

* Fulminant liver failure; or
* Concurrent (multi-organ transplant) or previous solid organ or bone marrow transplant; or
* Chronic renal dialysis at time of transplant; or
* Dependency on more than 1 inotropic agent to maintain hemodynamics; or
* Ventilator dependent at time of transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants in the OLP Registry will be all adult primary liver transplant candidates on the waiting list for liver transplant at a U.S. liver transplant center and who meet the eligibility criteria at the participating Registry centers.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patient Survival | 1 year post-Liver transplant
  1-year patient survival with the originally transplanted liver (patient and graft survival) post-Liver transplant.

OTHER OUTCOMES:
Safety Endpoint | 6 months post-Liver transplant
  6-months liver graft survival post-Liver transplant
Long Term Patient Survival | 2 years post-transplant
  K-M Patient survival at 1- and 2-years post-transplant
Long Term Graft Survival | 2 years post-transplant
  K-M Graft survival at 6 months, 1- and 2-years post-transplant

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Emory, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke Medical Center, Durham, North Carolina
  - Houston Methodist, Houston, Texas